CLINICAL TRIAL: NCT04937192
Title: SNP-based Prediction of Recurrence Risk in Kidney Stone Patients: a Prospective Multicenter Observational Study
Brief Title: SNP-based Prediction of Recurrence Risk in Kidney Stone Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Wuhan University Renmin Hospital (Unknown); The Second Affiliated Hospital of Kunming Medical University (Other); Tianjin Medical University Second Hospital (Other); Shenzhen People's Hospital (Other); 301 Hospital (Unknown); Zhongda Hospital (Other); People's Hospital of Xinjiang (Unknown); ZhuZhou Central Hospital (Other); Baoshan No.2 People's Hospital (Unknown); Guangdong No.2 People's Hospital (Unknown); Dehong People's Hospital (Unknown); Second Affiliated Hospital of Guangzhou Medical University (Other); Jiangmen Central Hospital (Other); Huizhou Municipal Central Hospital (Other); Yongzhou Center Hospital (Unknown); Longgang District People's Hospital of Shenzhen (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: MRER2013-001
Record Dates: First submitted 2021-06-10; First posted 2021-06-23 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Kidney Stone
Keywords: SNP; Kidney stone; Recurrence
MeSH Terms: conditions — Kidney Calculi; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood was obtained for DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney stone former
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this study is to gain new knowledge about genetic risk factors that may affect the kidney stone recurrence. The study seeks to understand if different forms of genes result in an increased risk of kidney stone recurrence.

DETAILED DESCRIPTION:
In this study, investigators are prospectively testing whether SNP are associated with kidney stone recurrence. Investigators will test the hypothesis that SNP predispose kidney stone patients to recurrence.

Investigators hope to identify predictors for the kidney stone recurrence. This would allow the identification of a subpopulation of kidney stone patients that would benefit most from prevention measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Kidney stone former who the stone was removed completely.
* Ability to give informed consent

Exclusion Criteria:

* Patient refuses or is unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney stone former who the stone was removed completely
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stone-free survival | From date of stone-free until the date of first stone recurrence (up to 7 years)
  Time to first stone recurrence from stone-free

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, M.D., Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided